CLINICAL TRIAL: NCT00226473
Title: Standard Palliative Care Versus Standard Palliative Care Plus Polychemotherapy (CVD-Protocol) in the Second-Line Therapy of Distant Metastasized Malignant Melanoma
Brief Title: Standard Palliative Care Versus Standard Palliative Care Plus Polychemotherapy in Metastasized Malignant Melanoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dermatologic Cooperative Oncology Group (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADO-MM-PAL8
Record Dates: First submitted 2005-09-25; First posted 2005-09-27 (Estimated); Last update posted 2006-06-21 (Estimated); Status verified 2005-09

CONDITIONS: Metastatic Melanoma
Keywords: malignant Melanoma; Chemotherapy; Metastasis; standard palliative care; best supportive care
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Cisplatin; Vindesine; Dacarbazine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Cisplatin, Vindesine, Dacarbazine (drugs)

SUMMARY:
The purpose of this multicenter study is to examine whether the proposed randomized treatment regime results in a significantly longer survival time and higher quality of life than any additionally applied multiple chemotherapy according to the CVD- scheme. So far neither established treatment regimes nor reliable data exist for the second-line chemotherapy of metastatic malignant melanoma. Patients are therefore mostly treated with single or multiple chemotherapeutics or/and immunomodulatory therapeutics. These regimes however imply often not only a higher toxicity but show rarely a response rate higher than 10%.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of metastatic melanoma (stage IV)
* progressive disease after first-line chemotherapy or immuno-chemotherapy
* Karnofsky-index > 60%
* informed consent

Exclusion Criteria:

* Uvea melanoma
* another primary malignancy except basal cell carcinoma or cervical carcinoma in situ
* severe and/or uncontrolled medical disease (diabetes mellitus, cardiac insufficiency)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Quality of life analysis
Objective tumor response rate in study arm B
Time to tumor progression
Cost analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ulrich, MD, Principal Investigator — Dept. of Dermatology, University Otto von Guericke, Leipziger Strasse 44, D-39120 Magdeburg, Germany; Axel Hauschild, MD, Principal Investigator — Dept. of Dermatology, University of Kiel, Schittenhelmstrasse 5, D-24105 Kiel, Germany; Peter Mohr, MD, Study Director — Dept. of Dermatology, Medical Center Buxtehude, Krankenhausstrasse 1, D-21614 Buxtehude, Germany
Locations (13):
- Germany (13):
  - Skin Cancer Unit, German Cancer Ressearch Center and Dept. of Dermatology, University Hospital of Mannheim, Mannheim, Baden-Wurttemberg
  - Dept. of Dermatology, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Dept. of Dermatology, University of Frankfurt, Frankfurt am Main, Hesse
  - Dept. of Dermatology, Medical Center Buxtehude, Buxtehude, Lower Saxony
  - Dept. of Dermatology, Hildesheim, Hildesheim, Lower Saxony
  - Dept. of. Dermatology, University of Saarland, Homburg, Homburg, Saaland
  - Dept. of Dermatology, University Otto von Guericke, Magdeburg, Saxony-Anhalt
  - Dept. of Dermatology, University of Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Dept. of Dermatology, University of Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Dept. of Dermatology, Charité Berlin, Berlin, State of Berlin
  - Dept. of Dermatology, Vivantes Clinics, Berlin, State of Berlin
  - Dept. of Dermatology, Helios Clinic Erfurt, Erfurt, Thuringia
  - Dept. of Dermatology, University of Jena, Jena, Thuringia

REFERENCES:
- [Background] Chapman PB, Einhorn LH, Meyers ML, Saxman S, Destro AN, Panageas KS, Begg CB, Agarwala SS, Schuchter LM, Ernstoff MS, Houghton AN, Kirkwood JM. Phase III multicenter randomized trial of the Dartmouth regimen versus dacarbazine in patients with metastatic melanoma. J Clin Oncol. 1999 Sep;17(9):2745-51. doi: 10.1200/JCO.1999.17.9.2745. PMID 10561349
- [Background] Creagan ET, Suman VJ, Dalton RJ, Pitot HC, Long HJ, Veeder MH, Vukov AM, Rowland KM, Krook JE, Michalak JC. Phase III clinical trial of the combination of cisplatin, dacarbazine, and carmustine with or without tamoxifen in patients with advanced malignant melanoma. J Clin Oncol. 1999 Jun;17(6):1884-90. doi: 10.1200/JCO.1999.17.6.1884. PMID 10561229
- [Background] Cure H, Souteyrand P, Ouabdesselam R, Roche H, Ravaud A, D'incan M, Viens P, Fargeot P, Lentz MA, Fumoleau P, Hanauske A, Chollet P. Results of a phase II trial with cystemustine at 90 mg/m(2) as a first- or second-line treatment in advanced malignant melanoma: a trial of the EORTC Clinical Studies Group. Melanoma Res. 1999 Dec;9(6):607-10. doi: 10.1097/00008390-199912000-00011. PMID 10661773
- [Background] Glimelius B, Ekstrom K, Hoffman K, Graf W, Sjoden PO, Haglund U, Svensson C, Enander LK, Linne T, Sellstrom H, Heuman R. Randomized comparison between chemotherapy plus best supportive care with best supportive care in advanced gastric cancer. Ann Oncol. 1997 Feb;8(2):163-8. doi: 10.1023/a:1008243606668. PMID 9093725
- [Background] Hauschild A, Garbe C, Stolz W, Ellwanger U, Seiter S, Dummer R, Ugurel S, Sebastian G, Nashan D, Linse R, Achtelik W, Mohr P, Kaufmann R, Fey M, Ulrich J, Tilgen W. Dacarbazine and interferon alpha with or without interleukin 2 in metastatic melanoma: a randomized phase III multicentre trial of the Dermatologic Cooperative Oncology Group (DeCOG). Br J Cancer. 2001 Apr 20;84(8):1036-42. doi: 10.1054/bjoc.2001.1731. PMID 11308250
- [Background] Propper DJ, Levitt NC, O'Byrne K, Braybrooke JP, Talbot DC, Ganesan TS, Thompson CH, Rajagopalan B, Littlewood TJ, Dixon RM, Harris AL. Phase II study of the oxygen saturation curve left shifting agent BW12C in combination with the hypoxia activated drug mitomycin C in advanced colorectal cancer. Br J Cancer. 2000 Jun;82(11):1776-82. doi: 10.1054/bjoc.2000.1138. PMID 10839290
- [Background] Thongprasert S, Sanguanmitra P, Juthapan W, Clinch J. Relationship between quality of life and clinical outcomes in advanced non-small cell lung cancer: best supportive care (BSC) versus BSC plus chemotherapy. Lung Cancer. 1999 Apr;24(1):17-24. doi: 10.1016/s0169-5002(99)00017-3. PMID 10403690